CLINICAL TRIAL: NCT04559854
Title: Mindful After Cancer Study: Fostering Positive Body Image, Sexual Health, and Well-being
Brief Title: Mindful After Cancer: A Mindfulness-based Therapy Intervention for Sexual Health After Cancer
Acronym: MAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Jessica Gorman, Associate Professor, Oregon State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-2019-003
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Gynecologic Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful After Cancer (Experimental): Participants will be asked to attend 8 weekly sessions via videoconference, and to complete home activities and mindfulness practice between sessions.
  Interventions: Behavioral: Mindful After Cancer

INTERVENTIONS:
Behavioral: Mindful After Cancer — The intervention includes eight weekly sessions (1.5-2 hours each), plus participant educational materials and audio recorded meditations, and is delivered to women in their homes via group videoconference led by a trained facilitator. Participants are asked to complete activities and mindfulness practice between sessions.

SUMMARY:
The objectives of this study are to: 1) adapt a mindfulness-based therapy program designed to help women manage their sexual and body image concerns after cancer (Mindful After Cancer, MAC) to a videoconference format and 2) assess the feasibility, acceptability, and preliminary effects of the program among breast and gynecologic cancer survivors.

DETAILED DESCRIPTION:
The specific aims are: 1) Assess the feasibility of the MAC program when delivered via videoconference and 2) Assess preliminary effects of the the program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast or gynecologic cancer at least one year prior to enrollment
* Completed primary cancer treatment
* English speaking
* Have access to a computer, smart phone, or tablet with internet access
* Ability to spend 15-30 minutes per day on program activities

Exclusion Criteria:

- Stage 0 (carcinoma in situ)

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 22 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Gorman, PhD, MPH, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindful After Cancer
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Education [Count of Participants; unit: Participants]
  College graduate | 20
  Did not graduate from college | 2
Income [Count of Participants; unit: Participants]
  < $50,000 annual income | 8
  > $50,000 annual income | 14
Employment Status [Count of Participants; unit: Participants]
  Employed | 15
  Unemployed | 7
Health Insurance Coverage [Count of Participants; unit: Participants]
  Yes | 22
  No | 0
Relationship status [Count of Participants; unit: Participants]
  Partnered | 15
  Not Partnered | 7
Sexual Orientation [Count of Participants; unit: Participants]
  Bisexual | 4
  Heterosexual | 18
Cancer Type [Count of Participants; unit: Participants]
  Breast | 21
  Ovarian | 1
Self-Reported Cancer Stage [Count of Participants; unit: Participants] — Based on self report only. Higher stage generally indicates a more advanced cancer.
  Participants
    I | 12
    II | 5
    III | 3
    IV | 1
    Unknown | 1
Age at Cancer Diagnosis [Mean (Standard Deviation); unit: years] | 47.0 (8.1)
Time Since Cancer Diagnosis [Mean (Standard Deviation); unit: years] | 6.0 (5.9)
Has Biological Child(ren) [Count of Participants; unit: Participants] | 15
Sexually Active [Count of Participants; unit: Participants] | 13
Current Contraception Use [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility/ Enrollment in the Study
Description: Percentage of participants enrolled of those eligible
Time Frame: Baseline (T1)
Measure: Number; unit: Percentage enrolled of eligible
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 22
Percentage enrolled of eligible | 78.6

2. Primary Outcome: Feasibility/ Retention in the Study
Description: Number and percentage of participants completing all assessments
Time Frame: 1 month post-intervention (T2)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 22
Participants | 22

3. Primary Outcome: Feasibility/ Retention in the Intervention
Description: Number and percentage attending at least 6 of 8 sessions
Time Frame: 1 month post-intervention (T2)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 22
Participants | 18

4. Primary Outcome: Acceptability of the Intervention
Description: Endorsement of 10 items characterizing acceptability of the intervention (e.g., the program met my expectations). Range 10-100. Higher score indicates better acceptability.
Time Frame: 1 month post-intervention (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 22
score on a scale | 75.5 (22.9)

5. Secondary Outcome: Change From Baseline Interest in Sexual Activity at 1 Month
Description: PROMIS Sexual Function and Satisfaction 2.0. 2 items. Range 2-10. Higher score indicates more interest in sexual activity.
Time Frame: Baseline (T1) and 1 month post-intervention (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 20
score on a scale
  T1 Mean, SD | 4.4 (1.4)
  T2 Mean, SD | 5.0 (1.7)

6. Secondary Outcome: Change From Baseline Satisfaction With Sex Life at 1 Month
Description: New Sexual Satisfaction Scale- Short Form (NSSS-S). 12 items. Range 12-60. Higher score indicates more sexual satisfaction.
Time Frame: Baseline (T1) and 1 month post-intervention (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 6
score on a scale
  T1 Mean, SD | 35 (6.8)
  T2 Mean, SD | 37.3 (7.4)

7. Secondary Outcome: Change From Baseline Self-efficacy at 1 Month
Description: Self-efficacy for Managing Chronic Disease Scale (adapted). 6 items. Range 6-60. Higher score indicates better self-efficacy for managing sexual health after cancer.
Time Frame: Baseline (T1) and 1 month post-intervention (T2)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 20
score on a scale | 0.06 [-0.87 to 0.98]

8. Secondary Outcome: Change From Baseline Body Image at 1 Month
Description: Body Image Scale. 10 items. Range 0-30. Higher score indicates poorer body image.
Time Frame: Baseline (T1) and 1 month post-intervention (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 21
score on a scale
  T1 Mean, SD | 15.2 (7.1)
  T2 Mean, SD | 13.1 (8.2)

9. Secondary Outcome: Change From Baseline Body Appreciation at 1 Month
Description: Body Appreciation Scale. 13 items. Range 13-65. Higher score indicates more positive body appreciation.
Time Frame: Baseline (T1) and 1 month post-intervention (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 21
score on a scale
  T1 Mean, SD | 3.2 (0.7)
  T2 Mean, SD | 3.6 (0.7)

10. Secondary Outcome: Change From Baseline Anxiety at 1 Month
Description: PROMIS Emotional Distress Anxiety Short Form 6a. 6 items. Range 6-30. Higher score indicates greater anxiety symptoms.
Time Frame: Baseline (T1) and 1 month post-intervention (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 21
score on a scale
  T1 Mean, SD | 15.0 (5.4)
  T2 Mean, SD | 12.9 (4.4)

11. Secondary Outcome: Change From Baseline Depression at 1 Month
Description: Center for Epidemiologic Studies Depression Scale (CES-D). 20 items. Range 0-60. Higher score indicates greater depressive symptoms
Time Frame: Baseline (T1) and 1 month post-intervention (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 20
score on a scale
  T1 Mean, SD | 16.3 (9.0)
  T2 Mean, SD | 13.9 (11.3)

12. Secondary Outcome: Change in Facets of Baseline Mindfulness at 1 Month
Description: Five-Facet Mindfulness Questionnaire (FFMQ-15). 15 items with 5 sub-scales: Observe, Describe; Act with Awareness; Non-Judgement, Non-Reactivity. Sub-scale score range 3-15. Higher score indicates greater mindfulness.
Time Frame: Baseline (T1) and 1 month post-intervention (T2)
Measure: Mean (Standard Deviation); unit: score on a subscale
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 20
score on a subscale
  Observe subscale T1 Mean, SD | 10.8 (2.1)
  Observe subscale T2 Mean, SD | 9.6 (0.9)
  Acting with Awareness subscale T1 Mean, SD | 9.3 (2.0)
  Acting with Awareness subscale T2 Mean, SD | 10.8 (2.2)
  Non-reactivity subscale T1 Mean, SD | 9.7 (2.4)
  Non-reactivity subscale T2 Mean, SD | 8.9 (1.0)
  Non-judging subscale T1 Mean, SD | 10.7 (2.4)
  Non-judging subscale T2 Mean, SD | 8.8 (1.4)
  Describing subscale T1 Mean, SD | 10.3 (2.4)
  Describing subscale T2 Mean, SD | 10.0 (1.5)

13. Secondary Outcome: Change From Baseline Self-compassion at 1 Month
Description: Self-Compassion Scale short form. 12 items. Total score is calculated based on mean of item responses (each item ranges 1-5). Higher mean score indicates greater self-compassion.
Time Frame: Baseline (T1) and 1 month post-intervention (T2)
Measure: Mean (Standard Deviation); unit: mean score on a scale
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 20
mean score on a scale
  T1 Mean, SD | 3.0 (0.7)
  T2 Mean, SD | 2.9 (0.2)

14. Secondary Outcome: Change From Baseline Relationship Quality at 1 Month
Description: Dyadic Adjustment Scale short form (DAS-7). Range 0-36. Higher score indicates more positive relationship quality
Time Frame: Baseline (T1) and 1 month post-intervention (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindful After Cancer
Number analyzed (Participants) | 14
score on a scale
  T1 Mean, SD | 24.0 (6.5)
  T2 Mean, SD | 25.3 (5.7)

ADVERSE EVENTS:
Time Frame: Duration of study, approximately 3-4 months
Arm/Group | Mindful After Cancer
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT04559854/Prot_SAP_000.pdf